CLINICAL TRIAL: NCT00462839
Title: The Accuracy of Blood Loss Estimation After Simulated Vaginal Delivery
Brief Title: Accuracy of Blood Loss Estimation After Vaginal Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Cynthia Wong, Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0524-029
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Results first posted 2011-12-09 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Postpartum Hemorrhage
Keywords: Estimated Blood Loss; Obstetrics; postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calibrated drapes viewed first (Experimental): Caregivers were shown calibrated drape demonstrating level of blood and asked to estimate amount of blood in collection bag. These same individuals were then crossed over and shown non-calibrated drapes and asked to estimate the amount of blood they contained.
  Interventions: Procedure: blood loss estimation
- Non-calibrated drapes viewed first (Active Comparator): Standard vaginal delivery drape (non-calibrated) was shown to caregiver who was asked to estimate amount of blood. These same individuals were then crossed over and shown calibrated delivery drapes and asked to estimate the amount of blood they contained.
  Interventions: Procedure: blood loss estimation

INTERVENTIONS:
Procedure: blood loss estimation — Participants were randomized in blocks, by provider type to view either the four calibrated stations or the four non-calibrated stations. The order of the volumes within each set of stations was randomized. Participants received a data card for each station on which they wrote the volume estimated. After each station, the data card was collected. Alterations to the estimations were not allowed once the answers were recorded. Subjects were then crossed over to the other group and asked to estimate the blood volumes in the non-calibrated drapes if they had first viewed the calibrated drape or the calibrated drape if they had viewed the non-calibrated drape. The order of viewing the four volumes was again randomized. The volumes were the same at the corresponding station for the calibrated and non-calibrated stations so the impact of the calibration markings on accuracy could be determined.
  Other Names: Estimated Blood Loss (EBL)

SUMMARY:
Post-partum hemorrhage (PPH) is defined as blood loss greater than 500 mL after vaginal delivery. Delayed diagnosis of PPH is a major cause of maternal morbidity and mortality. Obstetricians estimate blood loss at delivery by visual estimation of blood collected in the obstetric drapes. Blood is often mixed with urine and surgical sponges. The urine, blood, and sponges collect in a cone shaped plastic bag that is suspended from the perineum during delivery. Visual estimation of blood loss is insensitive in diagnosing PPH. In one study visual assessment of blood loss underestimated postpartum blood loss by 33% to 50% compared to an objective measurement of blood loss using photospectrometry. Other studies have shown that the magnitude of underestimation increases as the amount of blood loss is increased. A limitation of previous studies is that there is no "gold standard" for blood loss determination in the third stage of labor. Care providers (obstetricians, anesthesiologists, and labor & delivery nurses) need to be able to accurately estimate blood loss in order to better care for mothers and prevent morbidity and mortality. It is unknown whether provider type or experience (obstetric and anesthesiology resident, fellow, attending physicians, and nurses) influences the accuracy of blood loss estimation, or whether blood loss estimation can be improved by providing graduated markings on the vaginal delivery drape.

DETAILED DESCRIPTION:
Packed red blood cells discarded by the blood bank will be mixed with normal saline to simulate whole blood with a hematocrit of 33%. A total of eight isolated study stations will be set up (study participants will only be able to visualize the vaginal delivery drape for one station at a time). The simulated blood will be mixed with urine and sponges and be placed in suspended blood collection drapes which are used during vaginal deliveries at Northwestern Memorial Hospital. Two types of drapes will be used: drapes without calibrated markings and drapes with calibrated markings. Calibrated volume markings will begin at 500 mL at 500 mL intervals to 2500 mL.

Study participants will be randomized to one of two groups. Randomization will occur in blocks depending on provider type. Group 1 will view the unmarked vaginal collection drapes first and Group 2 will view the collection drapes with the calibrated markings first. Both groups will analyze the initial four study stations in random order. At the completion of the four study stations, the group which evaluated the drapes without markings will cross over to view the stations with calibrated markings and the group that views uncalibrated drapes will then view the calibrated drapes.

Each study participant will view a station and write his/her estimation of blood loss on a data card. Study participants will NOT be allowed to change answers once they have been recorded.

Demographic data on study participants will include provider type, level of training/years of practice, and gender.

ELIGIBILITY:
Inclusion Criteria:

* Any anesthesia or obstetric attending or resident may participate provided that they have rotated through obstetrics/obstetric anesthesia.

Exclusion Criteria:

* Any provider that does not complete all of the stations will be excluded from analysis. Any participant who chooses to withdraw from the study will also be excluded from the analysis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2006-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Wong, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] C. Beckman. Obstetrics and Gynecology. Post Partum Hemorrhage, Chapter 12. 3rd edition. Lippincott Williams & Wilkins 1998; 154-161.
- [Background] Cunningham FG, Leveno KL, Bloom SL, et al. Williams Obstetrics, 22th ed, New York: McGraw-Hill, 2005.
- [Background] Patel A, Goudar SS, Geller SE, Kodkany BS, Edlavitch SA, Wagh K, Patted SS, Naik VA, Moss N, Derman RJ. Drape estimation vs. visual assessment for estimating postpartum hemorrhage. Int J Gynaecol Obstet. 2006 Jun;93(3):220-4. doi: 10.1016/j.ijgo.2006.02.014. Epub 2006 Apr 12. PMID 16626718
- [Background] Prasertcharoensuk W, Swadpanich U, Lumbiganon P. Accuracy of the blood loss estimation in the third stage of labor. Int J Gynaecol Obstet. 2000 Oct;71(1):69-70. doi: 10.1016/s0020-7292(00)00294-0. No abstract available. PMID 11044547

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted on two separate dates at Prentice Women's Hospital. Eight stations were set up in 8-12 hour periods in an empty labor and delivery room. Participants were randomized in blocks by provider type. The order of the volumes was randomized. Subjects were not informed that the volumes in the two groups were the same.
Groups:
- Calibrated Vaginal Delivery Drapes Viewed First: Calibrated drapes had volume markings beginning at 500ml with 500ml increments to a total of 2500ml. Subjects were randomized to either view calibrated or uncalibrated (standard of care) drapes and asking to estimated volume of blood loss. Subjects were then crossed over and experiment repeated.
- Noncalibrated Drapes Viewed First: No distinguishable volume markings on drape (standard of care). Subjects were randomized to either view calibrated or uncalibrated (standard of care) drapes and asking to estimated volume of blood loss. Subjects were then crossed over and experiment repeated.
Period: Viewed First
Arm/Group | Calibrated Vaginal Delivery Drapes Viewed First | Noncalibrated Drapes Viewed First
Started | 53 | 53
Completed | 53 | 53
Not Completed | 0 | 0
Period: Viewed Second
Arm/Group | Calibrated Vaginal Delivery Drapes Viewed First | Noncalibrated Drapes Viewed First
Started | 53 | 53
Completed | 53 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calibrated Vaginal Delivery Drapes Viewed First | Noncalibrated Drapes Viewed First | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 53 | 106
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 32 | 66
  Male | 19 | 21 | 40
Region of Enrollment [Number; unit: participants]
  United States | 53 | 53 | 106

OUTCOME MEASURES:

1. Primary Outcome: Difference in Actual Blood Volume and Estimated Blood Volume in Milliliters.
Description: Two types of drapes were used: drapes with and without volume calibrations. Calibrated drapes had volume markings beginning at 500ml with 500ml increments to a total of 2500ml. The participants were asked to estimate the volume contained in the bag and the difference in milliliters between the estimate and actual volume was calculated.
Time Frame: 1 hour
Population: per protocal
Measure: Mean (95% Confidence Interval); unit: milliliters
Arm/Group | Calibrated Vaginal Delivery Drapes Viewed First | Noncalibrated Drapes Viewed First
Number analyzed (Participants) | 53 | 53
milliliters
  300 ml | -20.8 [-56.8 to 15.1] | -41.7 [-77.7 to -5.7]
  500 ml | -53.5 [-100.6 to -6.4] | -96.0 [-143.0 to -48.8]
  1000 ml | -32.8 [-150.3 to 84.6] | -145.3 [-262.8 to -27.8]
  2000 ml | -178 [-328.0 to -28.4] | -829.8 [-980.0 to -680.0]
Statistical Analysis 1: Comparison: Calibrated Vaginal Delivery Drapes Viewed First vs Noncalibrated Drapes Viewed First; Repeated measures ANOVA comparing all levels of blood estimation (P=0.0002). Post-hoc comparisons using Bonferroni corrects t-tests; Test type: Superiority or Other; p < 0.05, ANOVA — Post-hoc comparison of 500ml, 1000ml and 2000ml volumes were greater in the non-calibrated drape first group. Post-hoc comparisons made using Bonferroni correct t-test for 8 comparisons

2. Secondary Outcome: Number and Type of Care Providers Assigned to Study Arms.
Time Frame: 1 hour
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Calibrated Vaginal Delivery Drapes Viewed First | Noncalibrated Drapes Viewed First
Number analyzed (Participants) | 53 | 53
participants
  Anesthesia | 21 | 22
  Obstetrics | 20 | 22
  Nursing | 12 | 9
Statistical Analysis 1: Comparison: Calibrated Vaginal Delivery Drapes Viewed First vs Noncalibrated Drapes Viewed First; Test type: Superiority or Other; p = 0.76, Chi-squared, Corrected

3. Secondary Outcome: Level of Training
Time Frame: 1 hour
Measure: Number; unit: participants
Arm/Group | Calibrated Vaginal Delivery Drapes Viewed First | Noncalibrated Drapes Viewed First
Number analyzed (Participants) | 53 | 53
participants
  Attending physician | 19 | 22
  Resident physician | 22 | 22
  Nurse | 12 | 9
Statistical Analysis 1: Comparison: Calibrated Vaginal Delivery Drapes Viewed First vs Noncalibrated Drapes Viewed First; Test type: Superiority or Other; p = 0.72, Chi-squared, Corrected

4. Secondary Outcome: Number of Years of Clinical Experience Providing Patient Care Requiring Blood Loss Estimation.
Time Frame: 1 hour
Measure: Number; unit: participants
Arm/Group | Calibrated Vaginal Delivery Drapes Viewed First | Noncalibrated Drapes Viewed First
Number analyzed (Participants) | 53 | 53
participants
  < 5 years | 30 | 29
  5-10 years | 11 | 13
  > 10 years | 12 | 11
Statistical Analysis 1: Comparison: Calibrated Vaginal Delivery Drapes Viewed First vs Noncalibrated Drapes Viewed First; Test type: Superiority or Other; p = 0.89, Chi-squared, Corrected

ADVERSE EVENTS:
Arm/Group | Calibrated Vaginal Delivery Drapes Viewed First | Noncalibrated Drapes Viewed First
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 0/53 | 0/53

LIMITATIONS AND CAVEATS:
A limitation to our study is that we asked participants to estimate blood loss based on inspection of the conical drape only. We did not ask them to estimate blood loss in hidden places. In addition, this was not an actual delivery but a simulation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes